CLINICAL TRIAL: NCT00833326
Title: A Study of ARRY-334543 and Docetaxel in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Array Biopharma, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Array BioPharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARRAY-543-104
Record Dates: First submitted 2009-01-29; First posted 2009-02-02 (Estimated); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — ARRY-334543; Docetaxel; Antimitotic Agents; Injections, Subcutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ARRY-334543 + docetaxel + prophylactic growth factors (Experimental)
  Interventions: Drug: ARRY-334543, EGFR/ErbB2 inhibitor; oral; Drug: Docetaxel, mitotic inhibitor; intravenous; Drug: Prophylactic growth factors; subcutaneous

INTERVENTIONS:
Drug: ARRY-334543, EGFR/ErbB2 inhibitor; oral — multiple dose, escalating
Drug: Docetaxel, mitotic inhibitor; intravenous — multiple dose, single schedule
Drug: Prophylactic growth factors; subcutaneous — standard of care

SUMMARY:
This is a Phase 1 study during which patients with advanced/metastatic solid tumors will receive investigational study drug ARRY-334543 and docetaxel (with prophylactic growth factor support). Patients will receive increasing doses of study drug in combination with docetaxel in order to achieve the highest dose of study drug possible that will not cause unacceptable side effects. Patients will be followed to see what side effects the combination causes and what effectiveness the combination has, if any, in treating the cancer. Approximately 30 patients from the US will be enrolled in this study.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of any advanced/metastatic solid tumor suitable for treatment with docetaxel.
* Tumor recurred or progressed following at least one line of chemotherapy, except if no standard of care exists or if the patient refuses standard of care treatment.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1 or 2.
* Must be able to take and retain oral medications.
* Other criteria exist.

Key Exclusion Criteria:

* Active concomitant malignancies.
* Uncontrolled or symptomatic brain metastases (if a patient has brain metastases and is on steroids, the steroid dose must be stable for at least 30 days prior to study start).
* Known positive serology for the human immunodeficiency virus (HIV), hepatitis B and/or hepatitis C.
* Requiring intravenous (IV) alimentation.
* Pregnancy or lactation.
* Chemotherapy, anticancer immunotherapy, monoclonal antibodies or biologics within 21 days prior to first dose of study drug.
* Anti-ErbB1 and/or ErbB2 targeted therapy or anticancer hormonal therapy within 14 days prior to first dose of study drug.
* History of hypersensitivity to or intolerance of docetaxel.
* Other criteria exist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Establish the maximum tolerated dose (MTD) of study drug in combination with docetaxel. | Duration of study
Characterize the safety profile of study drug in combination with docetaxel in terms of adverse events, clinical laboratory tests and electrocardiograms. | Duration of study
Characterize the pharmacokinetics (PK) of study drug and docetaxel. | Duration of study

SECONDARY OUTCOMES:
Assess the efficacy of the study drug in combination with docetaxel in terms of tumor response. | Duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - Mayo Cancer Center, Rochester, Minnesota
  - Sarah Cannon Research Institute, Nashville, Tennessee